CLINICAL TRIAL: NCT02196012
Title: "The UTK Health Study" A Technology-Based Weight Loss Intervention for the Reduction of Overweight and Obesity Among College Students."
Brief Title: A Technology-Based Intervention for the Reduction of Overweight and Obesity Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9271B
Record Dates: First submitted 2014-04-28; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Overweight and Obesity
Keywords: overweight; obesity; Technology; College Students
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): The intervention condition will contain multiple components: nutrition education, physical activity, social support, social media (Pinterest and Facebook), and smartphone applications for self-monitoring. Students in this condition will have access to the private study website, which will be the central platform for delivery of the program materials and social support. The website, developed using Wordpress.com, will include nutrition materials, exercise videos, a forum, and links to the study's Facebook and Pinterest pages
  Interventions: Behavioral: Intervention group
- attention control condition (Active Comparator): Students randomized to the attention control condition will receive educational emails three times per week. Nutrition materials will be sent once a week, and links to the YouTube exercise videos will be sent twice a week. At the start of the program, students will be emailed a link to the Pandora workout station. The materials sent to the control group will be the same materials posted on the website for the intervention group. Participants will access the emailed lessons and videos each week at their own convenience. Individuals in the attention control condition will not have access to the study website or social media pages.
  Interventions: Behavioral: attention control condition

INTERVENTIONS:
Behavioral: Intervention group
  Arms: Lifestyle counseling
Behavioral: attention control condition
  Arms: attention control condition

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability and efficacy of a two month technology-based weight loss program for overweight and obese college students.

DETAILED DESCRIPTION:
A randomized controlled trial design will be employed to investigate the effectiveness, feasibility, and acceptability of a technology-based weight loss pilot intervention for the reduction of overweight and obesity in college students. Participants will be randomly assigned to one of two conditions: (1) 8-week intervention group, or (2) 8-week attention control group. Both conditions include 8 weekly lessons over 8 weeks. Undergraduate students (n=100) age 18-22 years who are overweight or obese (BMI ≥ 25 kg/m2) will be recruited from the University of Tennessee Knoxville. Measurements will be taken at baseline and 8 weeks. Since the study is a technology-based intervention, research staff will collect height and weight measures for BMI through a novel approach, utilizing Skype video conferencing.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility will include UTK undergraduate students who are overweight or obese (BMI ≥ 25 kg/m2) and between 18-22 years of age, with access to the Internet, a personal computer (laptop, tablet, or desktop computer), and a smartphone.

Exclusion Criteria:

* Any individual who does not meet all the inclusion criteria will be excluded from participation in the study.
* Students who have a medical condition that precludes adherence to dietary recommendations
* Who are currently prescribed medications that may impact weight, or who are currently participating in or planning to participate in another weight loss programs in the next six months
* Who have been diagnosed with a major psychiatric illness (e.g., bipolar disorder, schizophrenia, or depression) within the last 12 months
* Who are pregnant or plan to become pregnant in the next six months
* Who have given birth within the last six months
* Who have been diagnosed with any type of eating disorder within the past 12 months will be ineligible.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
body mass index (BMI) | 2 months

SECONDARY OUTCOMES:
feasibility | 2 months
  A mixed methods approach, including online surveys and focus groups, was employed to assess the feasibility of the pilot study. Feasibility was assessed through recruitment and retention data and self-reported records of participant engagement.

OTHER OUTCOMES:
acceptability | 2 months
  Participants in both groups completed an online post-intervention survey. Data were collected and compiled through SurveyMonkey. Surveys were comprised of a combination of closed-ended and open-ended questions. Participants completed text-based focus group using Skype group messaging. Participants were asked to provide feedback on each technology tool in the program, the website, methods of delivery, the duration of the program, and the overall program. A benefit was that the online tools allowed students to maintain anonymity, which could have encouraged participation and sharing.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States